CLINICAL TRIAL: NCT06203301
Title: The Relationships of Resistance Exercise, Walking, Myokine Secretion, Sarcopenia, Muscle Loss, Quality of Life, and Predictors in Cancer Patients Receiving Chemoradiotheray
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N202109030
Record Dates: First submitted 2023-12-18; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Walking

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (No Intervention): No exercise intervention measures will be implemented. The patient will carry out daily life according to his past living habits and continue to be followed for at least one year.
- resistance exercise group (Experimental): Resistance exercise training begins before the patient undergoes concurrent chemoradiotherapy, radiotherapy, or chemotherapy. The patients were given resistance exercise training for 45 minutes each time, 3 times a week, for 12 consecutive weeks. After that, the patient is asked to regularly perform resistance exercise for at least 1 year.
  Interventions: Behavioral: resistance exercise and walking
- walking group (Experimental): Walking training begins before the patient undergoes simultaneous radiochemotherapy, radiation therapy, or chemotherapy, and requires continuous walking for 15 minutes at least twice a day and at least 5 days a week. Or walk for at least 150 minutes a week and walk for at least 15 minutes continuously each time for 12 consecutive weeks of walking training. After that, ask the patient to walk regularly for at least 1 year.
  Interventions: Behavioral: resistance exercise and walking
- resistance exercise and walking group (Experimental): Before patients receive concurrent chemoradiotherapy, radiotherapy, or chemotherapy, they are given resistance exercise training and walking training for 12 consecutive weeks. After that, the patient is asked to regularly perform resistance exercise and walking for at least 1 year.
  Interventions: Behavioral: resistance exercise and walking

INTERVENTIONS:
Behavioral: resistance exercise and walking — After receiving the cases, they were divided into 4 groups by random allocation:
  1. Control group: No exercise intervention measures are performed, and the patients carry out their daily lives according to their past living habits.
  2. Resistance exercise group: Resistance exercise training begins before the patients receive simultaneous radiochemotherapy, radiation therapy, or chemotherapy. The patients are given resistance exercise training for 45 minutes each time, 3 times a week, for 12 consecutive weeks. Afterwards, the patient is asked to regularly perform resistance exercise on his own for at least 1 year.
  3. Walking group: Walking training begins before the patients receive simultaneous radiochemotherapy, radiation therapy, or chemotherapy. They should walk continuously for 15 minutes at least twice a day and continue walking at least 5 days a week. Or walk for at least 150 minutes a week and walk for at least 15 minutes continuously each time for 12 consecutive weeks of walk
  Arms: resistance exercise and walking group; resistance exercise group; walking group

SUMMARY:
Cancer is the first most common cause of death in Taiwan. The application of surgery and chemoradiotherapy are used for treatment of patients with cancer. However, loss of muscle mass, low muscle strength, low physical performance, and sarcopenia are induced during chemoradiotherapy, consequently increased the risk of hematological toxicity and nonhematological toxicity, decreased quality of life and survival rate. It was reported that skeletal muscle can secretion of myokines, which contribute to muscle synthesis, growth, repair, or atrophy. Investigators suggest that detection of blood concentration of myokines and sarcopenia-related predictors can early detection potential individuals who are susceptibility to sarcopenia in cervical cancer patients receiving chemoradiotherapy. Also, resistance exercise was demonstrated to improve muscle mass, muscle strength, physical performance, and sarcopenia. Investigators suggest that resistance exercise can prevent cervical cancer patients from sarcopenia and improve quality of life through regulation the concentration of myokines. However, there was no study has been investigated their relationships. Therefore, investigators will conduct a randomized controlled trial study to estimate (1) the effect of resistance exercise, walking on regulation myokine secretion, improving skeletal muscle mass, muscle strength, physical performance, sarcopenia, and quality of life in cancer receiving chemoradiotherapy; (2) myokine level, muscle mass, muscle strength, physical performance, and sarcopenia incidence in cancer patients before and after receiving chemoradiotherapy.

DETAILED DESCRIPTION:
Cancer is the first most common cause of death in Taiwan. The application of surgery and chemoradiotherapy are used for treatment of patients with cancer. However, loss of muscle mass, low muscle strength, low physical performance, and sarcopenia are induced during chemoradiotherapy, consequently increased the risk of hematological toxicity and nonhematological toxicity, decreased quality of life and survival rate. It was reported that skeletal muscle can secretion of myokines, which contribute to muscle synthesis, growth, repair, or atrophy. Investigators suggest that detection of blood concentration of myokines and sarcopenia-related predictors can early detection potential individuals who are susceptibility to sarcopenia in cervical cancer patients receiving chemoradiotherapy. Also, resistance exercise was demonstrated to improve muscle mass, muscle strength, physical performance, and sarcopenia. Investigators suggest that resistance exercise can prevent cervical cancer patients from sarcopenia and improve quality of life through regulation the concentration of myokines. However, there was no study has been investigated their relationships. Therefore, investigators will conduct a randomized controlled trial study to estimate (1) the effect of resistance exercise, walking on regulation myokine secretion, improving skeletal muscle mass, muscle strength, physical performance, sarcopenia, and quality of life in cancer receiving chemoradiotherapy; (2) myokine level, muscle mass, muscle strength, physical performance, and sarcopenia incidence in cancer patients before and after receiving chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients receiving chemoradiotherap
* age 20-70 years old
* participants who are available for doing resistance exercise and/or walking after physical assessment by physician
* education level >=elementary school

Exclusion Criteria:

* Participants can't speak Mandarin, Taiwanese, or Hakka language.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
physical functional performance | From enrollment to the end of treatment at 12 weeks, then follow up for 1 year.
  This study plans to use the 5-time stand-up-sit test to assess physical functional performance. Five stand-up and sit-down tests lasting more than or equal to 12 seconds indicate that the patient's physical function performance is reduced.During the measurement, the patient is asked to sit on a chair about 40cm above the ground. The back of the chair is against the wall. The patient is asked to sit down against the back of the chair. The patient is asked to stand up. The patient is asked to do his best to stand up and stand upright five times continuously and without interruption. Sit down, keeping your hands folded on your chest.During the test, the patient stood up once and was asked to count the sounds. The test ended when the patient stood up for the fifth time.
muscle strength | From enrollment to the end of treatment at 12 weeks, then follow up for 1 year.
  Measuring the patient's muscle strength with a handgrip dynamometer(Hand Grip Strength, EH101, CAMYR, Guangdong)
muscle mass | From enrollment to the end of treatment at 12 weeks, then follow up for 1 year.
  In order to avoid radiation exposure when patients undergo testing and to facilitate repeated measurements, this research plan will use the Bioelectrical Impedance Analyzer (BIA) Inbody S10 to detect the skeletal muscle mass of the limbs of patients. The bioelectrical impedance analyzer is currently a commonly used analyzer for clinical measurement of body composition, using microcurrent to measure the human body.
the incidence of sarcopenia | From enrollment to the end of treatment at 12 weeks, then follow up for 1 year.
  The assessment of sarcopenia in this study uses the Asian Working Group for Sarcopenia (AWGS) diagnostic criteria as the criteria for screening sarcopenia, including: (1) low muscle strength: handgrip strength <28 kg for men, women <18 kg; (2) low physical performance: 5 stand-up and sit-down tests greater than or equal to 12 seconds; (3) loss of appendicular skeletal muscle mass (ASM): bioelectrical impedance analysis (BIA) men <7.0kg/m2, women <5.7kg/m2.
  If the skeletal muscle mass of the limbs is reduced combined with weakened muscle strength or physical functional performance, it is called sarcopenia; if the skeletal muscle mass of the limbs is reduced, the muscle strength is weakened, and the physical functional performance is reduced at the same time, it is severe sarcopenia.
effectively improve their quality of life | From enrollment to the end of treatment at 12 weeks, then follow up for 1 year.
  This study uses the Functional Assessment of Cancer Therapy-General (FACT-G) to assess the quality of life of patients.
The concentration of muscle hormones in the blood of cancer patients undergoing treatment | From enrollment to the end of treatment at 12 weeks, then follow up for 1 year.
  The specimen is collected based on the principle of collecting 5 mL of venous blood. The blood is injected into a special biochemical test tube containing Lithium heparin, an anticoagulant, and mixed gently to avoid blood coagulation and hemolysis.
  Centrifuge at 3500 rpm for 10 minutes, and separate the upper plasma for detection of muscle hormones in the blood, including: myonectin, irisin, decorin, fibroblast growth factor-21, interleukin-15, interleukin-6, myostatin, osteonectin, and brain-derived hormones.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taipei Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No